CLINICAL TRIAL: NCT01807390
Title: Perspectives for Receiving Open Versus MIS (PROMIS) - Patients' Perspectives on Surgical Treatment of Lung and Esophageal Cancer
Brief Title: Perspectives of Receiving Open Versus Minimally Invasive Surgery
Acronym: PROMIS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20120321-01H
Record Dates: First submitted 2013-02-25; First posted 2013-03-08 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Lung Cancer; Esophageal Cancer
Keywords: Minimally invasive surgery; Patient perspectives; Lung cancer; Esophageal cancer; Pain
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will examine the perspectives of patients' undergoing surgery for lung or esophageal cancer. It will examine both pre-op and post-op patient perspectives and opinions regarding pain and surgical complications. This study will also assess a general health related quality of life pre-op and post-op. Additionally, it will examine the importance of receiving care close to home and their support system.

Hypotheses:

1. The data will allow investigators to better understand the willingness of patients to participate in prospective, randomized studies comparing minimally invasive and open thoracic surgery. Patients will not be willing to undergo randomization to an open versus minimally invasive surgical procedure.
2. The pain associated with Minimally Invasive Surgery (MIS) will be perceived and documented as lesser than open surgery.
3. Patients may be willing to accept a higher risk of complications or more post-operative pain if they were given the option to be cared for closer to their home.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are surgical candidates for lung or esophageal cancer (entered at pre-op time point)

Exclusion Criteria:

* Below 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the Ottawa Hospital General Campus who are surgical candidates for lung or esophageal cancer over the age of 18.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain perceptions | Baseline, 4 weeks and 6 months
  Patients will rate their perceptions of pain associated with surgery both pre-op and at 4 weeks and 6 months post-op.

SECONDARY OUTCOMES:
Change in general health related quality of life | Baseline, 4 weeks and 6 months
  Patients will rate their general health related quality of life at pre-op, and post-op (4 weeks and 6 months) time points.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Gilbert, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided